CLINICAL TRIAL: NCT01276522
Title: Efficacy and Safety of Canakinumab in Schnitzler Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-SS-Canakinumab
Record Dates: First submitted 2011-01-12; First posted 2011-01-13 (Estimated); Last update posted 2012-05-24 (Estimated); Status verified 2012-05

CONDITIONS: Schnitzler Syndrome
Keywords: Schnitzler syndrome; IL-1 beta; Canakinumab; Ilaris; Treatment; Efficacy; Safety
MeSH Terms: conditions — Schnitzler Syndrome | interventions — canakinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Canakinumab (Experimental): A 6-month open-label, single treatment arm study of canakinumab 150 or 300 mg (in case of insufficient response to 150 mg) subcutaneous injection once per month.
  Interventions: Drug: Canakinumab

INTERVENTIONS:
Drug: Canakinumab — Monthly subcutaneous injection with 150mg Canakinumab for 6 months
  Other Names: Ilaris

SUMMARY:
Schnitzler syndrome is a disabling inflammatory disease, characterized by chronic urticaria, fever, arthralgia, bone pain and gammopathy, which can so far only be effectively treated with anakinra, an interleukin-1 receptor antagonist. However, this drug is not registered for use in Schnitzler syndrome, and it needs to be injected daily, which is uncomfortable and unpractical. Therefore other treatments targeting IL-1 are needed. Canakinumab is a long-acting monoclonal antibody against IL-1β that has been registered for bimonthly use in the rare autoinflammatory disease Cryopyrin-associated periodic syndrome (CAPS). We hypothesize that it will be effective in Schnitzler syndrome too in view of clinical similarities to CAPS and the targeting of IL-1B, which is also blocked by anakinra (which blocks both IL-1B and IL-1A).

This is a 6-month open-label, single treatment arm study of canakinumab 150 or 300 mg (in case of insufficient response to 150 mg) subcutaneous injection once per month in patients with active Schnitzler syndrome, in which efficacy and safety will be assessed.

DETAILED DESCRIPTION:
More on Canakinumab:

Canakinumab is a high-affinity human monoclonal anti-human interleukin-1β (IL-1β)antibody of the IgG1/k isotype), developed for the treatment of IL-1β driven inflammatory diseases. Canakinumab binds human IL-1β and functionally neutralizes the bioactivity of this pro-inflammatory cytokine. IL-1β is produced mainly by mononuclear phagocytes in response to injury and infection and plays a dominant role in the pathobiology of autoinflammatory syndromes (e.g. Cryopyrin associated periodic syndrome, CAPS), systemic Juvenile Idiopathic Arthritis and gout. Canakinumab is expected to treat the signs and symptoms of inflammation and the underlying structural damage of disease. Canakinumab has been administered in clinical trials as an intravenous (i.v.) infusion or as a subcutaneous (sc) injection and has been approved under the trade name ILARIS® in the US for patients ≥ 4 years of age with CAPS and in the European Union and Switzerland for CAPS patients ≥ 4 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of Schnitzler syndrome as per criteria (ref 1).
* Patients that have been / are treated with Anakinra must have demonstrated a partial or complete clinical response with an associated normalization of their biomarkers of inflammation (CRP).
* Male and female patients at least 18 years of age at the time of the screening visit.
* Patient's informed consent.
* Negative QuantiFERON test or negative Purified Protein Derivative (PPD) test (< 5 mm induration) at screening or within 1 month prior to the screening visit, according to the national guidelines. Patients with a positive PPD test (≥ 5 mm induration) at screening may be enrolled only if they have either a negative chest x-ray or a negative QuantiFERON test (QFT-TB G In-Tube).
* Adequate contraception in premenopausal females

Exclusion Criteria:

* Pregnant or nursing (lactating) women
* History of being immunocompromised, including a positive HIV at screening (ELISA and Western blot).
* Serologic evidence of hepatitis B or C infection
* Live vaccinations within 3 months prior to the start of the trial, during the trial, and up to 3 months following the last dose
* History of significant medical conditions, which in the Investigator's opinion would exclude the patient from participating in this trial
* History of recurrent and/or evidence of active bacterial, fungal, or viral infection(s)
* Use of the following therapies:

  * Anakinra within 24 hours prior to Baseline visit XML File Identifier : tl8ybe8lI1o6DeawQocCBa8TF/w=
  * Corticosteroids (oral prednisone (or equivalent)) > 1.0 mg/kg/day (or greater than the maximum of 60 mg/day for children over 60 kg) within 3 days prior to the Baseline visit
  * Intra-articular, peri-articular or intramuscular corticosteroid injections within 4 weeks prior to the Baseline visit
  * Any other investigational biologics within 8 weeks prior to the Baseline visit
  * Any other investigational drugs, other than investigational biologic treatment, within 30 days (or 3 months for investigational monoclonal antibodies) or 5 half-lives prior to the Baseline visit, whichever is longer
* History of hypersensitivity to any of the study drugs or to drugs of similar chemical classes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2011-01; Primary Completion 2011-05 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Complete or clinical remission at Day 14. | Day 14

SECONDARY OUTCOMES:
Complete or clinical remission at Day 3 and Day 7 | Day 3 and day 7
The prevention of disease relapse in patients who demonstrated complete remission at Day 14 | Day 15 until end
The change in biomarkers (CRP and SAA) and clinical parameters (physician and patient global assessment of disease activity) during the treatment and follow-up periods | Whole study
Time to relapse after the last canakinumab dose | Month 6 - 9
Safety and tolerability as well as PK/PD/IG properties of canakinumab in the treatment of patients with Schnitzler syndrome. | Whole study
Changes in patient quality of life by using: Medical Outcome Short Form (36) Health Survey (SF-36®). | Whole study
Optimal canakinumab dose and frequency in patients with Schnitzler syndrome | Whole study

CONTACTS AND LOCATIONS:
Overall Officials: Anna Simon, MD PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands

REFERENCES:
- [Background] de Koning HD, Bodar EJ, van der Meer JW, Simon A; Schnitzler Syndrome Study Group. Schnitzler syndrome: beyond the case reports: review and follow-up of 94 patients with an emphasis on prognosis and treatment. Semin Arthritis Rheum. 2007 Dec;37(3):137-48. doi: 10.1016/j.semarthrit.2007.04.001. Epub 2007 Jun 21. PMID 17586002
- [Background] de Koning HD, Bodar EJ, Simon A, van der Hilst JC, Netea MG, van der Meer JW. Beneficial response to anakinra and thalidomide in Schnitzler's syndrome. Ann Rheum Dis. 2006 Apr;65(4):542-4. doi: 10.1136/ard.2005.045245. Epub 2005 Aug 11. PMID 16096327
- [Background] Ryan JG, de Koning HD, Beck LA, Booty MG, Kastner DL, Simon A. IL-1 blockade in Schnitzler syndrome: ex vivo findings correlate with clinical remission. J Allergy Clin Immunol. 2008 Jan;121(1):260-2. doi: 10.1016/j.jaci.2007.09.021. Epub 2007 Oct 22. No abstract available. PMID 17936890
- [Background] Schuster C, Kranke B, Aberer E, Arbab E, Sturm G, Aberer W. Schnitzler syndrome: response to anakinra in two cases and a review of the literature. Int J Dermatol. 2009 Nov;48(11):1190-4. doi: 10.1111/j.1365-4632.2009.04151.x. PMID 20064173
- [Background] Martinez-Taboada VM, Fontalba A, Blanco R, Fernandez-Luna JL. Successful treatment of refractory Schnitzler syndrome with anakinra: comment on the article by Hawkins et al. Arthritis Rheum. 2005 Jul;52(7):2226-7. doi: 10.1002/art.21101. No abstract available. PMID 15986356
- [Background] Lipsker D, Veran Y, Grunenberger F, Cribier B, Heid E, Grosshans E. The Schnitzler syndrome. Four new cases and review of the literature. Medicine (Baltimore). 2001 Jan;80(1):37-44. doi: 10.1097/00005792-200101000-00004. PMID 11204501
- [Background] Lachmann HJ, Kone-Paut I, Kuemmerle-Deschner JB, Leslie KS, Hachulla E, Quartier P, Gitton X, Widmer A, Patel N, Hawkins PN; Canakinumab in CAPS Study Group. Use of canakinumab in the cryopyrin-associated periodic syndrome. N Engl J Med. 2009 Jun 4;360(23):2416-25. doi: 10.1056/NEJMoa0810787. PMID 19494217
- [Background] Lachmann HJ, Lowe P, Felix SD, Rordorf C, Leslie K, Madhoo S, Wittkowski H, Bek S, Hartmann N, Bosset S, Hawkins PN, Jung T. In vivo regulation of interleukin 1beta in patients with cryopyrin-associated periodic syndromes. J Exp Med. 2009 May 11;206(5):1029-36. doi: 10.1084/jem.20082481. Epub 2009 Apr 13. PMID 19364880
- [Derived] de Koning HD, Schalkwijk J, van der Ven-Jongekrijg J, Stoffels M, van der Meer JW, Simon A. Sustained efficacy of the monoclonal anti-interleukin-1 beta antibody canakinumab in a 9-month trial in Schnitzler's syndrome. Ann Rheum Dis. 2013 Oct;72(10):1634-8. doi: 10.1136/annrheumdis-2012-202192. Epub 2012 Oct 19. PMID 23087179